CLINICAL TRIAL: NCT02564536
Title: A Pilot Study of Pacritinib in Combination With Low Dose Decitabine in Patients With Intermediate-High Risk Myelofibrosis or MPN/MDS Syndromes
Brief Title: Pacritinib in Combination With Low Dose Decitabine in Intermediate-High Risk Myelofibrosis or Myeloproliferative Neoplasm (MPN)/Myelodysplastic Syndrome (MDS)
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of funding following full FDA clinical hold
Sponsor: Washington University School of Medicine (Other)
Collaborators: CTI BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201510166
Record Dates: First submitted 2015-09-29; First posted 2015-09-30 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Chronic Myelomonocytic Leukemia; Juvenile Myelomonocytic Leukemia; Atypical Chronic Myeloid Leukemia; Myeloproliferative Neoplasm; Myelodysplastic Syndromes; Myelofibrosis
MeSH Terms: conditions — Leukemia, Myelomonocytic, Chronic; Leukemia, Myelomonocytic, Juvenile; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Myeloproliferative Disorders; Myelodysplastic Syndromes; Primary Myelofibrosis | interventions — 11-(2-pyrrolidin-1-ylethoxy)-14,19-dioxa-5,7,26-triazatetracyclo(19.3.1.1(2,6).1(8,12))heptacosa-1(25),2(26),3,5,8,10,12(27),16,21,23-decaene; Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Arm 1: Pacritinib and Decitabine (Experimental): * Patients will receive one cycle of single agent pacritinib.
  * Patients who tolerate single agent pacritinib will then receive up to 11 cycles of pacritinib and decitabine combination therapy.
  * Patients who do not tolerate single agent pacritinib (require dose interruption for more than 7 days before Cycle 2 Day 1) will be considered non-evaluable and replaced.
  * Pacritinib will be administered orally at a dose of 200 mg twice daily continuously for Days 1 through 28 of a 28-day cycle.
  * Decitabine will be administered as a subcutaneous injection in clinic on Days 1, 5, 8, 12, 15, 19, 22, and 26 of a 28-day cycle.
  * Patients may continue treatment for up to 12 cycles.
  Interventions: Drug: Pacritinib; Drug: Decitabine

INTERVENTIONS:
Drug: Pacritinib — -Patients should take pacritinib at approximately the same times every day with a glass of water, with or without food.
Drug: Decitabine — -From commercial stock

SUMMARY:
For the first 28 day cycle, all patients will be treated with single agent pacritinib at 200 mg twice daily. The investigators chose this starting dose based on the previous three phase I studies of pacritinib as a single agent which showed that the maximum tolerated dose (MTD) to be 500 mg, and subsequently, the dose of 400 mg daily was recommended for the phase II studies.

Recently, the results of the phase III PERSIST-1 trial comparing pacritinib to best available therapy (BAT) in patients with MF was reported at the 2015 American Society of Clinical Oncology (ASCO) annual meeting. Pacritinib was found to be significantly more effective than BAT at reducing spleen volume at 24 weeks of therapy and improving constitutional symptoms.

Low dose decitabine has demonstrated depletion of DNMT1 in normal hematopoietic stem cells (HSC) without cytotoxicity and subcutaneous (SC) instead of intravenous (IV) administration may avoid high peak levels that can cause apoptosis. Furthermore, the low toxicity associated with low dose decitabine would allow for more frequent (1 to 3 times weekly) administration of the drug which would catch more cells in S-phase via greater exposure time. Based on these findings, a starting dose of decitabine 5 mg/m2 SC twice weekly should be well tolerated and effective in patients with MF and MPN/MDS syndromes when combined with pacritinib 400 mg daily.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of:

  * Primary MF or post-PV/ET MF classified as high risk, intermediate-2 risk, or intermediate-1 risk who are unresponsive or unable to receive current therapy which may or may not include ruxolitinib OR
  * MPN/MDS Syndrome (chronic myelomonocytic leukemia [CMML], juvenile myelomonocytic leukemia [JMML], atypical chronic myeloid leukemia [aCML], or MDS/MPN unclassifiable)
* ECOG 0-3
* Required laboratory values:

  * Neutrophil count of ≥ 0.5 x 109/L
  * Bone marrow blood blast count < 20%
  * AST and ALT ≤ 3 x ULN (≤ 5 x ULN if liver is involved by extramedullary hematopoiesis as judged by the investigator or if related to iron chelator therapy that was started within the prior 60 days)
  * Total creatinine < 2.5mg/dL
  * Total bilirubin ≤ 2.0 x ULN
* Age ≥ 18 years old at enrollment.
* If female, must be:

  * postmenopausal for at least 1 year before the screening visit OR
  * surgically sterile OR
  * agreeable to practicing 2 effective methods of contraception prior to study entry, for the duration of study participation, and for 30 days after the last dose of study treatment.
* Able to swallow pills.
* If a sexually active heterosexual male, must be agreeable to practicing 2 effective methods of contraception prior to study entry, for the duration of study participation, and for 30 days after the last dose of study treatment.
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

* Prior treatment with more than two JAK2 inhibitors or with pacritinib
* Known positive status for human immunodeficiency virus (HIV)
* Chronic, active, or acute viral hepatitis A, B, or C infection, or a hepatitis B or C carrier
* Use of chemotherapy, biologic therapy, radiation therapy, erythropoietin or related erythropoiesis stimulating agents, or investigational therapy within 2 weeks of the first dose of study drug
* History of allogeneic stem cell transplant or transplant eligible
* Currently receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to pacritinib or other agents used in the study
* Ongoing gastrointestinal medical condition such as Crohn's disease, inflammatory bowel disease, chronic diarrhea, or chronic constipation that could interfere with absorption of oral medication
* Active bleeding that requires hospitalization during the screening period
* Cardiovascular disease, including recent history of or currently clinically symptomatic and uncontrolled congestive heart failure, arrhythmia, angina, QTc prolongation or other QTc risk factors, myocardial infarction. Patients with CTCAE grade 2 cardiac arrhythmias may be considered for inclusion if the arrhythmias are stable, asymptomatic, and unlikely to affect patient safety. Patients will e excluded if they have ongoing cardiac dysrhythmias of CTCAE grade ≥ 3, corrected QT interval (QTc) prolongation > 450 ms, or other factors that increase the risk for QT interval prolongation (e.g., heart failure, hypokalemia [defined as serum potassium < 3.0 mEq/L that is persistent and refractory to correction], or family history of long QT interval syndrome).
* Other malignancy requiring active treatment at time of study entry
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, or serious medical or psychiatric illness/social situations that would limit compliance with study requirements.
* Life expectancy < 6 months
* Pregnant and/or breastfeeding. Patient must have a negative pregnancy test within 14 days of study entry.
* Receiving treatment with any potent CYP3A4 inhibitors within 7 days of the first dose of study drug
* Patients with MF who are eligible for enrollment in the pacritinib "PERSIST-2" study at WUSM (NCT02055781) HRPO 201406075.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-06 (Estimated); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Safety of regimen as measured by adverse events | 30 days after completion of treatment (up to 1 year)
  The descriptions and grading for adverse events are found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0

SECONDARY OUTCOMES:
Rate of objective response as defined by the International Working Group-Myeloproliferative Neoplasms Research and Treatment (IWG-MRT) consensus | End of treatment (up to 48 weeks)
  Objective response is defined as CR (complete remission/response) + PR (partial remission/response) + CI (clinical improvement).
Rate of hematologic response | End of treatment (up to 48 weeks)
  -Anemia response
  Anemia response is only applicable for patients with baseline hemoglobin level less than 10g/dL for 8 weeks or more and requires:
  *≥2 g/dL increase in hemoglobin level
  *becoming transfusion-independent (no RBC transfusions in past 1 month)
  -Platelet response
  Platelet response is only applicable for patients with a baseline platelet count of less than 50 x 10^9/L for 8 weeks or more, and requires:
  * 100% increase in platelet count AND
  * An absolute platelet count of at least 50 x 10^9/L
Rate of symptom response as measured by the total symptom score (TSS) | End of treatment (up to 48 weeks)
  A ≥50% reduction in the myeloproliferative neoplasm symptom assessment total symptom score
Rate of spleen response | End of treatment (up to 48 weeks)
  * A baseline splenomegaly that is palpable at 5-10 cm below the left costal margin becomes not palpable OR
  * A baseline splenomegaly that is palpable > 10 cm below the left costal margin decreases by ≥50% OR
  * A baseline splenomegaly that is palpable < 5 cm below the left costal margin is not eligible for spleen response OR
  * MRI or CT shows ≥35% spleen volume reduction

CONTACTS AND LOCATIONS:
Overall Officials: Camille Abboud, M.D., Principal Investigator — Washington University School of Medicine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu